CLINICAL TRIAL: NCT03494985
Title: A Clinical Study to Evaluate the Efficacy of an Experimental Oralbalance Gel, Oral Rinse and Spray Versus Water
Brief Title: A Clinical Study to Evaluate the Efficacy of Three Dry Mouth Relief Products Versus Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202902; RH01986 (Other: GSK)
Record Dates: First submitted 2018-04-05; First posted 2018-04-11 (Actual); Results first posted 2018-07-18 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia | interventions — Water

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The examiner and site staff reviewing the efficacy assessments were blinded to the treatment allocation of participants. All other study personnel (study statistician, data management staff and other employees of the Sponsor who may influence study outcomes) were blinded to the study treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OralBalance moisturizing gel (Experimental): All the participants in this arm used an experimental Oralbalance gel as instructed under the supervision of trained site staff on their visits.
  Interventions: Device: Experimental Oralbalance Moisturizing Gel
- Oral rinse (Experimental): All the participants in this arm used an Oral rinse as instructed under the supervision of trained site staff on their visits.
  Interventions: Device: Biotene Original Oral Rinse
- Moisturizing mouth spray (Experimental): All the participants in this arm used a moisturising mouth spray as instructed under the supervision of trained site staff on their visits.
  Interventions: Device: Biotene Moisturizing Mouth Spray
- Water only use (Sham Comparator): All the participants in this arm used water as instructed under the supervision of trained site staff on their visits.
  Interventions: Other: Water

INTERVENTIONS:
Device: Experimental Oralbalance Moisturizing Gel — Participants placed approximately a half inch length of the gel onto the tongue and spread thoroughly using their tongue. Participants used their assigned treatment products for 28 days as specified on their diary/instructions, at least twice and no more than 5 times daily.
  Arms: OralBalance moisturizing gel
Device: Biotene Original Oral Rinse — Participants rinsed their mouth with 15 milliliters (mL) of oral rinse for 30 seconds and spat out. Participants used their assigned treatment products for 28 days as specified on their diary/instructions, at least twice and no more than 5 times daily.
  Arms: Oral rinse
Device: Biotene Moisturizing Mouth Spray — Participants sprayed one jet directly into their mouth. Participants used their assigned treatment products for 28 days as specified on their diary/instructions, at least twice and no more than 5 times daily.
  Arms: Moisturizing mouth spray
Other: Water — Participants were allowed to take only one measured sip of water (15 mL) 30 minutes before the supervised product use. After the supervised treatment at the site, participants assigned to the water only treatment were allowed to sip water as often as required.
  Arms: Water only use

SUMMARY:
This study assessed the efficacy of three dry mouth products (including an experimental Oralbalance gel, oral rinse, and moisturizing spray) to relieve the feeling of dry mouth compared to water, in dry mouth population over a period of 28 days.

DETAILED DESCRIPTION:
This was a multi-centered (two-sites), examiner-blinded, four treatment arms, stratified (by Modified Dry Mouth Inventory [DMI] score), randomized, parallel group study in participants with self-reported dry mouth symptoms as determined by participant responses to the DMI. Participants used their assigned dry mouth treatment at home for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: a) No clinically significant and relevant abnormalities of medical history or oral examination., b) Absence of any condition that would impact on the subject's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements. Subjects with stable and controlled medical conditions with no overt medical conditions which would contraindicate participation (in the opinion of the Investigator or medically qualified designee) which would interfere with the conduct of the study.
* Self reported feeling of a dry mouth according to the modified DMI questions. Subject must answer at least 3 out of 5 questions with 'agree a little', 'agree' or 'strongly agree'.

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
* Previous participation in this study.
* Recent history (within the last 1 year) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family.
* Subject works in one of the following: Advertising, Journalism, Public Relations, Manufacturing, retail or distribution of medicines, medical devices or healthcare products, Market Research or Marketing.
* Use of prescription systemic parasympathetic medications (e.g. Pilocarpine), for the treatment of the feeling of dry mouth.
* At the discretion of the examiner, subjects currently under the care of a dental/medical professional specifically for the treatment of dry mouth.
* Evidence of gross intra-oral neglect or need for extensive dental therapy.
* Denture wearer (partial or complete dentures).
* Subject with dental implants.
* Subjects with untreated oral mucosal disease which in the opinion of the investigator could interfere with the study (e.g. current oral ulceration).
* Subject is currently undergoing radiotherapy and/or chemotherapy treatment.
* Any condition the investigator identifies that can confound the subject's ability to properly participate in the study e.g. Alzheimer's Disease.

Ages: 35 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2013-09-17 (Actual); Primary Completion 2014-01-10 (Actual); Study Completion 2014-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2 sites in United States of America.
Pre-assignment Details: 467 participants were screened, out of which 45 were not randomized to the study. 15 did not meet study criteria, 8 were lost to follow-up, 19 withdrew their consent, and 3 were due to other reason (not specified). 422 were enrolled in the study out of which 26 did not meet eligibility criteria. Remaining 396 started the study.
Period: Overall Study
Arm/Group | OralBalance Moisturizing Gel | Oral Rinse | Moisturizing Mouth Spray | Water Only Use
Started | 101 | 98 | 98 | 99
Completed | 96 | 92 | 92 | 94
Not Completed | 5 | 6 | 6 | 5
Not completed — Adverse Event | 3 | 2 | 3 | 0
Not completed — Other (Withdrawal of consent) | 2 | 3 | 2 | 5
Not completed — Other (Not specified) | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OralBalance Moisturizing Gel | Oral Rinse | Moisturizing Mouth Spray | Water Only Use | Total
Number analyzed (Participants) | 101 | 98 | 98 | 99 | 396
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 56.2 (10.19) | 52.6 (10.87) | 54.0 (9.80) | 52.7 (9.61) | 53.9 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 74 | 79 | 78 | 304
  Male | 28 | 24 | 19 | 21 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 11 | 7 | 16 | 40
  Not Hispanic or Latino | 95 | 87 | 91 | 83 | 356
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 2
  Asian | 2 | 1 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 17 | 16 | 13 | 59
  White | 85 | 77 | 80 | 84 | 326
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Modified Product Performance and Attributes Questionnaire I (PPAQ I) (Question Number 1: Relieving the Discomfort of Dry Mouth)
Description: Participants were asked to use the following scale to rate question 1 (Relieving the discomfort of dry mouth) of PPAQ I as it applied to the study product: 1= poor, 2= fair, 3= good, 4= very good, and 5= excellent. PPAQ I was assessed at 2 hours after supervised product use on Day 29 of treatment.
Time Frame: At Day 29 of treatment (2 hours after supervised product use)
Population: Intent to treat (ITT, N= 396) population defined as all randomized participants with at least one post-baseline assessment of efficacy. The ITT population was analyzed as per randomized treatment. Number of participants analyzed for this endpoint were part of the IIT population, evaluated on Day 29.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | OralBalance Moisturizing Gel | Oral Rinse | Moisturizing Mouth Spray | Water Only Use
Number analyzed (Participants) | 95 | 92 | 91 | 92
Score on scale | 2.7 (1.07) | 2.9 (0.99) | 2.6 (1.02) | 2.0 (0.95)
Statistical Analysis 1: Comparison: OralBalance Moisturizing Gel vs Water Only Use; Test type: Other; p < 0.0001, ANOVA — p-value was adjusted using Dunnett's method for multiple comparisons; ANOVA model with factors for treatment, study site and DMI stratification (mild, moderate, severe); Least square mean difference = 0.6, 95% CI 2-sided [0.4 to 0.9] — First named treatment minus second named treatment such that a positive value favours the first named treatment
Statistical Analysis 2: Comparison: Oral Rinse vs Water Only Use; Test type: Other; p < 0.0001, ANOVA — p-value was adjusted using Dunnett's method for multiple comparisons; ANOVA model with factors for treatment, study site and DMI stratification (mild, moderate, severe); LS mean difference = 0.9, 95% CI 2-sided [0.6 to 1.2] — First named treatment minus second named treatment such that a positive value favours the first named treatment
Statistical Analysis 3: Comparison: Moisturizing Mouth Spray vs Water Only Use; Test type: Other; p < 0.0001, ANOVA — p-value was adjusted using Dunnett's method for multiple comparisons; ANOVA model with factors for treatment, study site and DMI stratification (mild, moderate, severe); LS mean difference = 0.6, 95% CI 2-sided [0.3 to 0.9] — First named treatment minus second named treatment such that a positive value favours the first named treatment

2. Secondary Outcome: Modified Product Performance and Attributes Questionnaire I (PPAQ I) (Question Number 1:Relieving the Discomfort of Dry Mouth ) at Day 29
Description: Participants were asked to use the following scale to rate question 1 (Relieving the discomfort of dry mouth) of PPAQ I as it applied to the study product:1= poor, 2= fair, 3= good, 4= very good, and 5= excellent. PPAQ I was assessed at 30 minutes, 1 hour, and 4 hours after supervised product use on Day 29 of treatment.
Time Frame: At Day 29 of treatment (30 minutes, 1 hour and 4 hours after supervised product use)
Population: ITT (N= 396) population defined as all randomized participants with at least one post-baseline assessment of efficacy. The ITT population was analyzed as per randomized treatment.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | OralBalance Moisturizing Gel | Oral Rinse | Moisturizing Mouth Spray | Water Only Use
Number analyzed (Participants) | 101 | 98 | 98 | 99
Score on scale
  At 30 mins: number analyzed (Participants) | 94 | 92 | 91 | 92
  At 30 mins | 3.0 (0.94) | 3.2 (0.86) | 3.1 (1.00) | 2.3 (0.97)
  At 1 hour: number analyzed (Participants) | 93 | 92 | 91 | 92
  At 1 hour | 2.9 (0.97) | 3.2 (0.82) | 2.9 (0.97) | 2.2 (0.95)
  At 4 hours: number analyzed (Participants) | 95 | 92 | 90 | 93
  At 4 hours | 2.5 (1.11) | 2.7 (1.03) | 2.5 (1.02) | 1.9 (0.95)

3. Secondary Outcome: Modified Product Performance and Attributes Questionnaire I (PPAQ I) Question Number 1: Relieving the Discomfort of Dry Mouth) Day 1
Description: Participants were asked to use the following scale to rate question 1 (Relieving the discomfort of dry mouth) of PPAQ I as it applied to the study product: 1= poor, 2= fair, 3= good, 4= very good, and 5= excellent. PPAQ I was assessed at 30 minutes, 1 hour, 2, and 4 hours after supervised product use on Day 1 of treatment.
Time Frame: At Day 1 of treatment (30 minutes, 1 hour, 2 and 4 hours after supervised product use)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | OralBalance Moisturizing Gel | Oral Rinse | Moisturizing Mouth Spray | Water Only Use
Number analyzed (Participants) | 101 | 98 | 98 | 99
Score on scale
  At 30 minutes: number analyzed (Participants) | 96 | 94 | 95 | 94
  At 30 minutes | 2.8 (0.97) | 2.8 (0.81) | 2.7 (0.97) | 2.2 (0.97)
  At 1 hour: number analyzed (Participants) | 98 | 96 | 93 | 94
  At 1 hour | 2.8 (0.89) | 2.7 (0.81) | 2.7 (0.95) | 2.0 (0.94)
  At 2 hours: number analyzed (Participants) | 98 | 98 | 94 | 94
  At 2 hours | 2.6 (0.97) | 2.4 (0.89) | 2.5 (0.97) | 1.8 (0.86)
  At 4 hours: number analyzed (Participants) | 97 | 97 | 95 | 96
  At 4 hours | 2.4 (1.09) | 2.3 (1.06) | 2.3 (1.02) | 1.6 (0.88)

4. Secondary Outcome: Individual Scores of All Question From 2-12 of Modified Product Performance and Attributes Questionnaire I (PPAQ I)
Description: Participants were asked to use the following scale to rate question (Q) 2 to 12 of PPAQ I as it applied to the study product: 1= poor, 2= fair, 3= good, 4= very good, and 5= excellent. PPAQ I had following questions Q2: Feeling comfortable in the mouth, Q3: Soothing your mouth, Q4: Allowing you to speak without difficulty, Q5: Effectively moistens your mouth, Q6: Effectively lubricates your mouth, Q7: Helping to freshen your breath, Q8: Protecting your mouth from drying out, Q9: Providing whole mouth comfort, Q10: Helping you to swallow without difficulty, Q11: Helping mouth feel 'normal', Q12: Having a cooling sensation. PPAQ I was assessed at 30 minutes, 1 hour, 2, and 4 hours after supervised product use on Day 1 and 29 of treatment. Individual score for each question at different tome point was reported for this endpoint.
Time Frame: At Day 1 and 29 (30 minutes, 1 hour, 2 and 4 hours after supervised product use)
Population: ITT(N= 396) population defined as all randomized participants with at least one post-baseline assessment of efficacy. The ITT population was analyzed as per randomized treatment.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | OralBalance Moisturizing Gel | Oral Rinse | Moisturizing Mouth Spray | Water Only Use
Number analyzed (Participants) | 101 | 98 | 98 | 99
Score on scale
  Q2 at Day 1, 30 minutes: number analyzed (Participants) | 99 | 96 | 97 | 98
  Q2 at Day 1, 30 minutes | 3.1 (0.92) | 3.0 (0.79) | 2.9 (1.00) | 2.5 (1.10)
  Q2 at Day 1, 1 hour: number analyzed (Participants) | 98 | 97 | 98 | 97
  Q2 at Day 1, 1 hour | 2.9 (0.93) | 2.8 (0.82) | 2.8 (1.00) | 2.2 (1.03)
  Q2 at Day 1, 2 hours: number analyzed (Participants) | 98 | 98 | 98 | 96
  Q2 at Day 1, 2 hours | 2.7 (0.97) | 2.5 (0.93) | 2.6 (0.99) | 2.0 (0.95)
  Q2 at Day 1, 4 hours: number analyzed (Participants) | 98 | 98 | 97 | 97
  Q2 at Day 1, 4 hours | 2.4 (1.09) | 2.4 (1.05) | 2.4 (1.03) | 1.8 (0.94)
  Q2 at Day 29, 30 minutes: number analyzed (Participants) | 96 | 92 | 93 | 93
  Q2 at Day 29, 30 minutes | 3.0 (1.00) | 3.3 (0.85) | 3.2 (1.07) | 2.4 (0.97)
  Q2 at Day 29, 1 hour: number analyzed (Participants) | 95 | 92 | 92 | 93
  Q2 at Day 29, 1 hour | 3.0 (0.87) | 3.2 (0.85) | 3.0 (1.00) | 2.3 (1.03)
  Q2 at Day 29. 2 hours: number analyzed (Participants) | 96 | 92 | 92 | 91
  Q2 at Day 29. 2 hours | 2.7 (1.04) | 3.0 (0.93) | 2.8 (0.99) | 2.2 (1.01)
  Q2 at Day 29, 4 hours: number analyzed (Participants) | 96 | 92 | 91 | 92
  Q2 at Day 29, 4 hours | 2.7 (1.06) | 2.8 (1.00) | 2.6 (1.07) | 2.0 (0.99)
  Q3 at Day 1, 30 minutes: number analyzed (Participants) | 99 | 97 | 96 | 95
  Q3 at Day 1, 30 minutes | 3.1 (0.97) | 3.0 (0.82) | 2.8 (1.02) | 2.3 (1.05)
  Q3 at Day 1, 1 hour: number analyzed (Participants) | 98 | 97 | 96 | 95
  Q3 at Day 1, 1 hour | 2.8 (1.01) | 2.7 (0.78) | 2.7 (0.93) | 2.1 (1.07)
  Q3 at Day 1, 2 hours: number analyzed (Participants) | 98 | 97 | 96 | 93
  Q3 at Day 1, 2 hours | 2.6 (1.00) | 2.4 (0.91) | 2.5 (0.98) | 1.9 (0.93)
  Q3 at Day 1, 4 hours: number analyzed (Participants) | 95 | 97 | 96 | 94
  Q3 at Day 1, 4 hours | 2.3 (1.11) | 2.2 (1.00) | 2.3 (1.05) | 1.6 (0.86)
  Q3 at Day 29, 30 minutes: number analyzed (Participants) | 96 | 92 | 92 | 92
  Q3 at Day 29, 30 minutes | 3.0 (0.98) | 3.3 (0.87) | 3.1 (1.02) | 2.3 (0.99)
  Q3 at Day 29, 1 hour: number analyzed (Participants) | 96 | 92 | 92 | 91
  Q3 at Day 29, 1 hour | 2.8 (1.01) | 3.2 (0.86) | 3.0 (1.04) | 2.2 (1.01)
  Q3 at Day 29. 2 hours: number analyzed (Participants) | 96 | 92 | 92 | 92
  Q3 at Day 29. 2 hours | 2.7 (1.08) | 2.9 (0.97) | 2.7 (1.06) | 2.0 (1.02)
  Q3 at Day 29, 4 hours: number analyzed (Participants) | 96 | 92 | 91 | 90
  Q3 at Day 29, 4 hours | 2.6 (1.04) | 2.6 (1.01) | 2.5 (1.08) | 2.0 (1.05)
  Q4 at Day 1, 30 minutes: number analyzed (Participants) | 93 | 94 | 94 | 89
  Q4 at Day 1, 30 minutes | 3.6 (0.88) | 3.4 (0.83) | 3.4 (0.94) | 3.0 (1.12)
  Q4 at Day 1, 1 hour: number analyzed (Participants) | 91 | 90 | 94 | 85
  Q4 at Day 1, 1 hour | 3.3 (0.95) | 3.2 (0.75) | 3.1 (0.95) | 2.6 (1.05)
  Q4 at Day 1, 2 hours: number analyzed (Participants) | 91 | 90 | 94 | 88
  Q4 at Day 1, 2 hours | 3.1 (0.93) | 2.9 (0.83) | 2.9 (0.88) | 2.4 (1.00)
  Q4 at Day 1, 4 hours: number analyzed (Participants) | 88 | 90 | 94 | 88
  Q4 at Day 1, 4 hours | 2.9 (0.91) | 2.8 (0.92) | 2.8 (1.00) | 2.3 (0.99)
  Q4 at Day 29, 30 minutes: number analyzed (Participants) | 88 | 86 | 91 | 88
  Q4 at Day 29, 30 minutes | 3.3 (0.81) | 3.5 (0.84) | 3.4 (0.97) | 2.7 (1.02)
  Q4 at Day 29, 1 hour: number analyzed (Participants) | 86 | 85 | 91 | 84
  Q4 at Day 29, 1 hour | 3.2 (0.87) | 3.4 (0.78) | 3.2 (0.95) | 2.6 (0.99)
  Q4 at Day 29. 2 hours: number analyzed (Participants) | 86 | 85 | 89 | 85
  Q4 at Day 29. 2 hours | 3.1 (0.91) | 3.3 (0.87) | 3.0 (1.02) | 2.5 (0.97)
  Q4 at Day 29, 4 hours: number analyzed (Participants) | 87 | 85 | 89 | 86
  Q4 at Day 29, 4 hours | 3.0 (1.02) | 3.0 (0.90) | 2.7 (1.01) | 2.3 (1.04)
  Q5 at Day 1, 30 minutes: number analyzed (Participants) | 101 | 97 | 97 | 96
  Q5 at Day 1, 30 minutes | 3.1 (1.08) | 3.0 (0.92) | 3.0 (1.13) | 2.5 (1.13)
  Q5 at Day 1, 1 hour: number analyzed (Participants) | 99 | 97 | 96 | 96
  Q5 at Day 1, 1 hour | 2.8 (1.00) | 2.8 (0.83) | 2.9 (1.08) | 2.1 (1.11)
  Q5 at Day 1, 2 hours: number analyzed (Participants) | 98 | 98 | 97 | 96
  Q5 at Day 1, 2 hours | 2.6 (1.07) | 2.4 (0.93) | 2.5 (1.02) | 1.9 (1.06)
  Q5 at Day 1, 4 hours: number analyzed (Participants) | 97 | 98 | 97 | 96
  Q5 at Day 1, 4 hours | 2.3 (1.10) | 2.2 (1.04) | 2.2 (1.10) | 1.6 (0.91)
  Q5 at Day 29, 30 minutes: number analyzed (Participants) | 95 | 92 | 92 | 90
  Q5 at Day 29, 30 minutes | 3.1 (0.95) | 3.3 (0.93) | 3.1 (1.03) | 2.4 (1.00)
  Q5 at Day 29, 1 hour: number analyzed (Participants) | 95 | 92 | 92 | 91
  Q5 at Day 29, 1 hour | 2.9 (1.09) | 3.1 (0.92) | 2.9 (1.04) | 2.2 (1.06)
  Q5 at Day 29. 2 hours: number analyzed (Participants) | 95 | 92 | 92 | 92
  Q5 at Day 29. 2 hours | 2.7 (1.06) | 2.9 (0.94) | 2.7 (1.10) | 2.1 (1.00)
  Q5 at Day 29, 4 hours: number analyzed (Participants) | 95 | 92 | 91 | 91
  Q5 at Day 29, 4 hours | 2.6 (1.10) | 2.6 (0.98) | 2.4 (1.09) | 2.0 (1.00)
  Q6 at Day 1, 30 minutes: number analyzed (Participants) | 100 | 97 | 97 | 96
  Q6 at Day 1, 30 minutes | 3.1 (1.06) | 3.0 (0.86) | 2.9 (1.12) | 2.4 (1.18)
  Q6 at Day 1, 1 hour: number analyzed (Participants) | 98 | 98 | 96 | 94
  Q6 at Day 1, 1 hour | 2.8 (1.06) | 2.7 (0.89) | 2.8 (1.09) | 2.0 (1.06)
  Q6 at Day 1, 2 hours: number analyzed (Participants) | 98 | 97 | 97 | 95
  Q6 at Day 1, 2 hours | 2.6 (1.02) | 2.4 (0.94) | 2.4 (1.05) | 1.8 (0.98)
  Q6 at Day 1, 4 hours: number analyzed (Participants) | 97 | 97 | 97 | 96
  Q6 at Day 1, 4 hours | 2.2 (1.08) | 2.2 (1.05) | 2.1 (1.07) | 1.6 (0.86)
  Q6 at Day 29, 30 minutes: number analyzed (Participants) | 95 | 91 | 93 | 91
  Q6 at Day 29, 30 minutes | 3.1 (1.01) | 3.3 (0.92) | 3.1 (1.07) | 2.3 (1.04)
  Q6 at Day 29, 1 hour: number analyzed (Participants) | 96 | 91 | 92 | 90
  Q6 at Day 29, 1 hour | 2.9 (1.09) | 3.0 (0.94) | 3.0 (1.04) | 2.2 (1.04)
  Q6 at Day 29. 2 hours: number analyzed (Participants) | 95 | 91 | 92 | 92
  Q6 at Day 29. 2 hours | 2.7 (1.08) | 2.9 (0.94) | 2.7 (1.10) | 2.0 (0.99)
  Q6 at Day 29, 4 hours: number analyzed (Participants) | 96 | 91 | 91 | 90
  Q6 at Day 29, 4 hours | 2.6 (1.14) | 2.5 (0.97) | 2.4 (1.09) | 2.0 (0.98)
  Q7 at Day 1, 30 minutes: number analyzed (Participants) | 93 | 95 | 93 | 81
  Q7 at Day 1, 30 minutes | 2.8 (1.02) | 3.3 (0.92) | 3.2 (1.10) | 1.8 (1.06)
  Q7 at Day 1, 1 hour: number analyzed (Participants) | 88 | 95 | 93 | 74
  Q7 at Day 1, 1 hour | 2.5 (0.99) | 2.9 (0.80) | 2.7 (1.02) | 1.7 (1.06)
  Q7 at Day 1, 2 hours: number analyzed (Participants) | 87 | 95 | 90 | 70
  Q7 at Day 1, 2 hours | 2.4 (1.12) | 2.4 (0.85) | 2.4 (1.04) | 1.6 (0.91)
  Q7 at Day 1, 4 hours: number analyzed (Participants) | 85 | 95 | 90 | 72
  Q7 at Day 1, 4 hours | 2.1 (1.02) | 2.2 (0.98) | 2.1 (1.06) | 1.5 (0.89)
  Q7 at Day 29, 30 minutes: number analyzed (Participants) | 85 | 88 | 91 | 79
  Q7 at Day 29, 30 minutes | 2.8 (1.12) | 3.2 (0.84) | 3.0 (1.16) | 2.0 (1.04)
  Q7 at Day 29, 1 hour: number analyzed (Participants) | 84 | 89 | 90 | 79
  Q7 at Day 29, 1 hour | 2.7 (1.19) | 3.0 (0.89) | 2.7 (1.08) | 1.9 (1.03)
  Q7 at Day 29. 2 hours: number analyzed (Participants) | 83 | 88 | 90 | 78
  Q7 at Day 29. 2 hours | 2.5 (1.18) | 2.7 (1.03) | 2.4 (1.13) | 1.8 (0.98)
  Q7 at Day 29. 4 hours: number analyzed (Participants) | 83 | 88 | 90 | 79
  Q7 at Day 29. 4 hours | 2.4 (1.20) | 2.5 (1.11) | 2.2 (1.12) | 1.7 (0.91)
  Q8 at Day 1, 30 minutes: number analyzed (Participants) | 99 | 94 | 94 | 97
  Q8 at Day 1, 30 minutes | 2.8 (0.99) | 3.0 (0.92) | 2.9 (1.18) | 2.2 (1.12)
  Q8 at Day 1, 1 hour: number analyzed (Participants) | 98 | 97 | 95 | 96
  Q8 at Day 1, 1 hour | 2.8 (1.00) | 2.7 (0.88) | 2.6 (1.01) | 2.0 (1.08)
  Q8 at Day 1, 2 hours: number analyzed (Participants) | 98 | 95 | 96 | 95
  Q8 at Day 1, 2 hours | 2.5 (1.13) | 2.3 (0.93) | 2.4 (0.97) | 1.7 (0.90)
  Q8 at Day 1, 4 hours: number analyzed (Participants) | 97 | 96 | 96 | 97
  Q8 at Day 1, 4 hours | 2.2 (1.07) | 2.2 (1.06) | 2.2 (1.04) | 1.6 (0.94)
  Q8 at Day 29, 30 minutes: number analyzed (Participants) | 95 | 92 | 92 | 91
  Q8 at Day 29, 30 minutes | 3.0 (1.00) | 3.3 (0.95) | 3.0 (1.09) | 2.2 (0.98)
  Q8 at Day 29, 1 hour: number analyzed (Participants) | 95 | 91 | 92 | 92
  Q8 at Day 29, 1 hour | 2.9 (1.05) | 3.1 (0.94) | 2.8 (1.11) | 2.1 (1.03)
  Q8 at Day 29. 2 hours: number analyzed (Participants) | 95 | 92 | 92 | 92
  Q8 at Day 29. 2 hours | 2.6 (1.04) | 2.9 (0.99) | 2.6 (1.06) | 2.0 (0.97)
  Q8 at Day 29. 4 hours: number analyzed (Participants) | 95 | 91 | 91 | 92
  Q8 at Day 29. 4 hours | 2.5 (1.09) | 2.6 (1.02) | 2.3 (1.13) | 2.0 (1.02)
  Q9 at Day 1, 30 minutes: number analyzed (Participants) | 100 | 97 | 96 | 95
  Q9 at Day 1, 30 minutes | 3.0 (0.96) | 3.1 (0.84) | 2.9 (1.13) | 2.3 (1.10)
  Q9 at Day 1, 1 hour: number analyzed (Participants) | 97 | 94 | 96 | 95
  Q9 at Day 1, 1 hour | 2.8 (0.92) | 2.8 (0.80) | 2.7 (1.01) | 2.1 (1.04)
  Q9 at Day 1, 2 hours: number analyzed (Participants) | 98 | 97 | 95 | 96
  Q9 at Day 1, 2 hours | 2.6 (1.01) | 2.5 (0.87) | 2.5 (1.00) | 1.9 (0.95)
  Q9 at Day 1, 4 hours: number analyzed (Participants) | 97 | 94 | 95 | 97
  Q9 at Day 1, 4 hours | 2.4 (1.11) | 2.3 (1.04) | 2.2 (0.98) | 1.7 (0.85)
  Q9 at Day 29, 30 minutes: number analyzed (Participants) | 96 | 92 | 92 | 91
  Q9 at Day 29, 30 minutes | 3.0 (1.05) | 3.3 (0.90) | 3.1 (1.03) | 2.3 (1.03)
  Q9 at Day 29, 1 hour: number analyzed (Participants) | 95 | 92 | 92 | 92
  Q9 at Day 29, 1 hour | 2.9 (1.03) | 3.1 (0.90) | 3.0 (1.02) | 2.3 (1.01)
  Q9 at Day 29. 2 hours: number analyzed (Participants) | 95 | 92 | 92 | 92
  Q9 at Day 29. 2 hours | 2.6 (1.07) | 2.9 (0.93) | 2.7 (1.07) | 2.0 (0.98)
  Q9 at Day 29. 4 hours: number analyzed (Participants) | 95 | 92 | 91 | 92
  Q9 at Day 29. 4 hours | 2.6 (1.11) | 2.7 (0.96) | 2.4 (1.07) | 2.0 (1.01)
  Q10 at Day 1, 30 minutes: number analyzed (Participants) | 92 | 89 | 94 | 92
  Q10 at Day 1, 30 minutes | 3.1 (0.95) | 3.2 (0.85) | 3.1 (1.07) | 2.6 (1.18)
  Q10 at Day 1, 1 hour: number analyzed (Participants) | 89 | 89 | 94 | 96
  Q10 at Day 1, 1 hour | 2.9 (0.92) | 3.0 (0.74) | 3.0 (0.96) | 2.3 (1.03)
  Q10 at Day 1, 2 hours: number analyzed (Participants) | 90 | 90 | 93 | 94
  Q10 at Day 1, 2 hours | 2.8 (1.05) | 2.7 (0.86) | 2.7 (0.93) | 2.2 (1.00)
  Q10 at Day 1, 4 hours: number analyzed (Participants) | 87 | 90 | 93 | 94
  Q10 at Day 1, 4 hours | 2.8 (0.99) | 2.6 (1.05) | 2.5 (1.08) | 2.1 (1.05)
  Q10 at Day 29, 30 minutes: number analyzed (Participants) | 87 | 85 | 91 | 89
  Q10 at Day 29, 30 minutes | 3.2 (0.92) | 3.5 (0.81) | 3.2 (1.02) | 2.4 (0.99)
  Q10 at Day 29, 1 hour: number analyzed (Participants) | 87 | 85 | 90 | 88
  Q10 at Day 29, 1 hour | 3.0 (1.01) | 3.3 (0.79) | 3.0 (0.99) | 2.4 (0.94)
  Q10 at Day 29. 2 hours: number analyzed (Participants) | 85 | 85 | 91 | 87
  Q10 at Day 29. 2 hours | 2.9 (1.05) | 3.1 (0.83) | 2.8 (1.02) | 2.3 (0.95)
  Q10 at Day 29. 4 hours: number analyzed (Participants) | 86 | 84 | 89 | 89
  Q10 at Day 29. 4 hours | 2.8 (1.08) | 2.9 (0.92) | 2.7 (1.03) | 2.2 (1.02)
  Q11 at Day 1, 30 minutes: number analyzed (Participants) | 99 | 96 | 95 | 97
  Q11 at Day 1, 30 minutes | 3.0 (0.91) | 3.1 (0.94) | 3.1 (1.08) | 2.4 (1.18)
  Q11 at Day 1, 1 hour: number analyzed (Participants) | 98 | 97 | 96 | 97
  Q11 at Day 1, 1 hour | 2.8 (0.91) | 2.9 (0.89) | 2.8 (1.06) | 2.2 (1.01)
  Q11 at Day 1, 2 hours: number analyzed (Participants) | 98 | 97 | 96 | 98
  Q11 at Day 1, 2 hours | 2.6 (1.01) | 2.6 (0.92) | 2.4 (0.98) | 2.0 (1.02)
  Q11 at Day 1, 4 hours: number analyzed (Participants) | 95 | 96 | 96 | 99
  Q11 at Day 1, 4 hours | 2.5 (1.09) | 2.4 (1.05) | 2.3 (1.05) | 1.9 (0.96)
  Q11 at Day 29, 30 minutes: number analyzed (Participants) | 95 | 92 | 92 | 92
  Q11 at Day 29, 30 minutes | 3.1 (0.97) | 3.3 (0.94) | 3.2 (0.99) | 2.4 (1.03)
  Q11 at Day 29, 1 hour: number analyzed (Participants) | 96 | 92 | 92 | 91
  Q11 at Day 29, 1 hour | 2.9 (0.92) | 3.1 (0.90) | 3.0 (0.98) | 2.3 (1.01)
  Q11 at Day 29, 2 hours: number analyzed (Participants) | 95 | 92 | 92 | 92
  Q11 at Day 29, 2 hours | 2.7 (0.99) | 2.9 (0.94) | 2.7 (1.06) | 2.1 (0.96)
  Q11 at Day 29. 4 hours: number analyzed (Participants) | 95 | 92 | 91 | 91
  Q11 at Day 29. 4 hours | 2.6 (1.05) | 2.7 (0.94) | 2.5 (1.09) | 2.1 (0.97)
  Q12 at Day 1, 30 minutes: number analyzed (Participants) | 93 | 93 | 92 | 84
  Q12 at Day 1, 30 minutes | 2.6 (1.16) | 3.1 (1.01) | 2.9 (1.21) | 2.2 (1.25)
  Q12 at Day 1, 1 hour: number analyzed (Participants) | 88 | 94 | 90 | 78
  Q12 at Day 1, 1 hour | 2.3 (1.12) | 2.7 (1.01) | 2.5 (1.03) | 2.0 (1.26)
  Q12 at Day 1, 2 hours: number analyzed (Participants) | 88 | 94 | 86 | 76
  Q12 at Day 1, 2 hours | 2.2 (1.07) | 2.1 (0.91) | 2.1 (0.99) | 1.7 (0.94)
  Q12 at Day 1, 4 hours: number analyzed (Participants) | 87 | 93 | 85 | 75
  Q12 at Day 1, 4 hours | 1.9 (0.96) | 2.0 (0.97) | 2.0 (0.92) | 1.6 (0.93)
  Q12 at Day 29, 30 minutes: number analyzed (Participants) | 84 | 89 | 88 | 83
  Q12 at Day 29, 30 minutes | 2.8 (1.12) | 3.1 (0.96) | 2.9 (1.10) | 2.1 (0.98)
  Q12 at Day 29, 1 hour: number analyzed (Participants) | 85 | 88 | 88 | 80
  Q12 at Day 29, 1 hour | 2.5 (1.11) | 2.8 (0.97) | 2.6 (1.11) | 2.0 (0.95)
  Q12 at Day 29. 2 hours: number analyzed (Participants) | 86 | 86 | 86 | 81
  Q12 at Day 29. 2 hours | 2.3 (1.12) | 2.6 (0.99) | 2.3 (1.15) | 1.7 (0.87)
  Q12 at Day 29. 4 hours: number analyzed (Participants) | 85 | 87 | 86 | 80
  Q12 at Day 29. 4 hours | 2.3 (1.18) | 2.3 (1.06) | 2.1 (1.07) | 1.7 (0.91)

5. Secondary Outcome: Individual Scores for All Questions of Modified Product Performance and Attributes Questionnaire I (PPAQ I) at Day 8
Description: Participants were asked to use the following scale to rate questions of PPAQ I as it applied to the study product: 1= poor, 2= fair, 3= good, 4= very good, and 5= excellent. PPAQI had following questions Q1: Relieving the discomfort of dry mouth Q2: Feeling comfortable in the mouth, Q3: Soothing your mouth, Q4: Allowing you to speak without difficulty, Q5: Effectively moistens your mouth, Q6: Effectively lubricates your mouth, Q7: Helping to freshen your breath, Q8: Protecting your mouth from drying out, Q9: Providing whole mouth comfort, Q10: Helping you to swallow without difficulty, Q11: Helping mouth feel 'normal', Q12: Having a cooling sensation. PPAQ I was assessed at 2 hours after supervised product use on Day 8 of treatment.
Time Frame: At Day 8 (2 hours after supervised product use)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | OralBalance Moisturizing Gel | Oral Rinse | Moisturizing Mouth Spray | Water Only Use
Number analyzed (Participants) | 101 | 98 | 98 | 99
Score on scale
  Q1 at Day 8, 2 hours: number analyzed (Participants) | 97 | 93 | 95 | 93
  Q1 at Day 8, 2 hours | 2.8 (0.98) | 3.0 (0.86) | 2.9 (0.86) | 2.1 (0.92)
  Q2 at Day 8, 2 hours: number analyzed (Participants) | 96 | 93 | 96 | 94
  Q2 at Day 8, 2 hours | 2.9 (0.97) | 3.0 (0.79) | 3.0 (1.00) | 2.2 (0.98)
  Q3 at Day 8, 2 hours: number analyzed (Participants) | 96 | 93 | 94 | 91
  Q3 at Day 8, 2 hours | 2.8 (1.04) | 2.9 (0.76) | 2.8 (0.97) | 2.0 (0.92)
  Q4 at Day 8, 2 hours: number analyzed (Participants) | 87 | 87 | 93 | 89
  Q4 at Day 8, 2 hours | 3.3 (0.89) | 3.2 (0.75) | 3.2 (0.97) | 2.5 (1.00)
  Q5 at Day 8, 2 hours: number analyzed (Participants) | 96 | 93 | 94 | 94
  Q5 at Day 8, 2 hours | 2.8 (1.00) | 3.0 (0.93) | 2.9 (1.07) | 2.1 (1.04)
  Q6 at Day 8, 2 hours: number analyzed (Participants) | 96 | 93 | 94 | 90
  Q6 at Day 8, 2 hours | 2.8 (0.98) | 2.9 (0.90) | 2.8 (1.11) | 2.0 (1.09)
  Q7 at Day 8, 2 hours: number analyzed (Participants) | 85 | 90 | 93 | 76
  Q7 at Day 8, 2 hours | 2.6 (1.09) | 2.9 (0.84) | 2.6 (1.02) | 1.5 (0.84)
  Q8 at Day 8, 2 hours: number analyzed (Participants) | 96 | 93 | 95 | 94
  Q8 at Day 8, 2 hours | 2.7 (1.00) | 2.9 (0.90) | 2.7 (1.07) | 1.9 (0.94)
  Q9 at Day 8, 2 hours: number analyzed (Participants) | 97 | 93 | 95 | 94
  Q9 at Day 8, 2 hours | 2.8 (0.97) | 2.9 (0.81) | 2.8 (1.07) | 2.1 (0.98)
  Q10 at Day 8, 2 hours: number analyzed (Participants) | 86 | 86 | 93 | 88
  Q10 at Day 8, 2 hours | 3.0 (0.92) | 3.2 (0.77) | 3.0 (0.99) | 2.4 (1.01)
  Q11 at Day 8, 2 hours: number analyzed (Participants) | 96 | 93 | 94 | 94
  Q11 at Day 8, 2 hours | 2.9 (0.90) | 3.0 (0.81) | 2.8 (1.02) | 2.1 (1.02)
  Q12 at Day 8, 2 hours: number analyzed (Participants) | 87 | 90 | 88 | 81
  Q12 at Day 8, 2 hours | 2.3 (1.10) | 2.7 (0.84) | 2.4 (1.03) | 1.7 (0.91)

6. Secondary Outcome: Individual Questions Scores of Modified Product Performance and Attributes Questionnaire II (PPAQ II)
Description: Participants were asked to use the following scale to rate questions of PPAQ II as it applied to the study product: 1= poor, 2= fair, 3= good, 4= very good, and 5= excellent. PPAQ II had following questions; Q1: Providing relief all night, Q2: Reducing the number of times you wake up from dry mouth, Q3: Feeling less parched when you wake up, Q4: Having a long lasting dry mouth relief, Q5. Having a long lasting lubricating effect, Q6: Having a long lasting moisturizing effect. PPAQ II was assessed before supervised product use on Day 8 and 29 of treatment.
Time Frame: At Day 8 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | OralBalance Moisturizing Gel | Oral Rinse | Moisturizing Mouth Spray | Water Only Use
Number analyzed (Participants) | 101 | 98 | 98 | 99
Score on scale
  Q1 at Day 8: number analyzed (Participants) | 94 | 91 | 95 | 90
  Q1 at Day 8 | 2.5 (0.96) | 2.7 (0.93) | 2.6 (1.00) | 2.2 (0.91)
  Q1 at Day 29: number analyzed (Participants) | 94 | 88 | 90 | 84
  Q1 at Day 29 | 2.7 (1.11) | 3.0 (0.93) | 2.8 (1.18) | 2.2 (1.08)
  Q2 at Day 8: number analyzed (Participants) | 89 | 82 | 87 | 88
  Q2 at Day 8 | 2.7 (0.95) | 2.9 (0.83) | 2.8 (0.94) | 2.1 (0.95)
  Q2 at Day 29: number analyzed (Participants) | 84 | 82 | 84 | 86
  Q2 at Day 29 | 3.1 (1.06) | 3.2 (0.96) | 2.9 (1.18) | 2.3 (1.20)
  Q3 at Day 8: number analyzed (Participants) | 95 | 91 | 94 | 92
  Q3 at Day 8 | 2.5 (0.94) | 2.8 (0.90) | 2.6 (0.99) | 1.9 (1.02)
  Q3 at Day 29: number analyzed (Participants) | 95 | 91 | 91 | 88
  Q3 at Day 29 | 2.7 (1.09) | 3.0 (1.08) | 2.6 (1.18) | 2.1 (1.12)
  Q4 at Day 8: number analyzed (Participants) | 97 | 93 | 95 | 94
  Q4 at Day 8 | 2.6 (0.97) | 2.7 (0.89) | 2.6 (0.98) | 1.9 (0.90)
  Q4 at Day 29: number analyzed (Participants) | 96 | 90 | 93 | 88
  Q4 at Day 29 | 2.8 (1.15) | 3.1 (1.07) | 2.8 (1.07) | 2.2 (1.08)
  Q5 at Day 8: number analyzed (Participants) | 96 | 93 | 93 | 90
  Q5 at Day 8 | 2.6 (0.98) | 2.8 (0.93) | 2.5 (1.00) | 1.9 (0.91)
  Q5 at Day 29: number analyzed (Participants) | 96 | 90 | 92 | 88
  Q5 at Day 29 | 2.8 (1.11) | 3.0 (1.06) | 2.8 (1.11) | 2.0 (1.06)
  Q6 at Day 8: number analyzed (Participants) | 96 | 93 | 94 | 90
  Q6 at Day 8 | 2.6 (1.00) | 2.8 (0.94) | 2.5 (0.92) | 1.9 (1.00)
  Q6 at Day 29: number analyzed (Participants) | 96 | 90 | 91 | 85
  Q6 at Day 29 | 2.8 (1.15) | 3.0 (1.08) | 2.8 (1.12) | 2.1 (1.11)

7. Secondary Outcome: Area Under Curve (AUC) up to 4 Hours After Treatment- Response of All Question of the Modified Product Performance and Attributes Questionnaire I (PPAQ I)
Description: The AUC was calculated for the interval starting at the time of the 30 minute response and ending at the time of the last valid reading using the trapezoidal method on Day 1 and Day 29. AUC was calculated for the score of the individual question of PPAQ1. All the questions were scored using the following scale: 1= poor, 2= fair, 3= good, 4= very good, and 5= excellent.
Time Frame: At Day 1 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on scale/seconds
Arm/Group | OralBalance Moisturizing Gel | Oral Rinse | Moisturizing Mouth Spray | Water Only Use
Number analyzed (Participants) | 101 | 98 | 98 | 99
Scores on scale/seconds
  Q1, AUC At Day 1: number analyzed (Participants) | 93 | 94 | 92 | 90
  Q1, AUC At Day 1 | 2.6 (0.88) | 2.5 (0.79) | 2.5 (0.85) | 1.9 (0.79)
  Q1, AUC At Day 29: number analyzed (Participants) | 93 | 92 | 90 | 92
  Q1, AUC At Day 29 | 2.7 (0.96) | 2.9 (0.88) | 2.7 (0.93) | 2.0 (0.89)
  Q2, AUC At Day 1: number analyzed (Participants) | 95 | 96 | 96 | 95
  Q2, AUC At Day 1 | 2.7 (0.88) | 2.6 (0.80) | 2.6 (0.83) | 2.0 (0.87)
  Q2, AUC At Day 29: number analyzed (Participants) | 95 | 92 | 91 | 91
  Q2, AUC At Day 29 | 2.8 (0.93) | 3.0 (0.85) | 2.8 (0.92) | 2.2 (0.95)
  Q3, AUC At Day 1: number analyzed (Participants) | 94 | 97 | 95 | 91
  Q3, AUC At Day 1 | 2.6 (0.93) | 2.5 (0.75) | 2.5 (0.86) | 1.9 (0.85)
  Q3, AUC At Day 29: number analyzed (Participants) | 96 | 92 | 91 | 90
  Q3, AUC At Day 29 | 2.7 (0.97) | 2.9 (0.86) | 2.7 (0.94) | 2.1 (0.96)
  Q4, AUC At Day 1: number analyzed (Participants) | 87 | 90 | 91 | 81
  Q4, AUC At Day 1 | 3.1 (0.78) | 3.0 (0.73) | 2.9 (0.78) | 2.5 (0.95)
  Q4, AUC At Day 29: number analyzed (Participants) | 85 | 85 | 87 | 83
  Q4, AUC At Day 29 | 3.1 (0.85) | 3.2 (0.79) | 3.0 (0.88) | 2.5 (0.95)
  Q5, AUC At Day 1: number analyzed (Participants) | 96 | 97 | 96 | 94
  Q5, AUC At Day 1 | 2.6 (0.94) | 2.5 (0.79) | 2.5 (0.93) | 1.9 (0.91)
  Q5, AUC At Day 29: number analyzed (Participants) | 94 | 92 | 91 | 90
  Q5, AUC At Day 29 | 2.7 (0.99) | 2.9 (0.86) | 2.7 (0.98) | 2.1 (0.95)
  Q6, AUC At Day 1: number analyzed (Participants) | 95 | 97 | 96 | 92
  Q6, AUC At Day 1 | 2.6 (0.90) | 2.4 (0.80) | 2.5 (0.93) | 1.8 (0.88)
  Q6, AUC At Day 29: number analyzed (Participants) | 95 | 91 | 91 | 88
  Q6, AUC At Day 29 | 2.8 (1.01) | 2.9 (0.86) | 2.7 (0.98) | 2.1 (0.93)
  Q7, AUC At Day 1: number analyzed (Participants) | 81 | 94 | 86 | 65
  Q7, AUC At Day 1 | 2.4 (0.94) | 2.5 (0.75) | 2.5 (0.93) | 1.6 (0.93)
  Q7, AUC At Day 29: number analyzed (Participants) | 82 | 87 | 87 | 73
  Q7, AUC At Day 29 | 2.6 (1.10) | 2.8 (0.92) | 2.5 (1.03) | 1.8 (0.94)
  Q8, AUC At Day 1: number analyzed (Participants) | 95 | 92 | 92 | 92
  Q8, AUC At Day 1 | 2.5 (0.94) | 2.4 (0.80) | 2.4 (0.87) | 1.8 (0.86)
  Q8, AUC At Day 29: number analyzed (Participants) | 95 | 91 | 91 | 91
  Q8, AUC At Day 29 | 2.7 (0.98) | 2.9 (0.89) | 2.6 (0.98) | 2.0 (0.94)
  Q9, AUC At Day 1: number analyzed (Participants) | 95 | 93 | 94 | 93
  Q9, AUC At Day 1 | 2.6 (0.88) | 2.6 (0.75) | 2.5 (0.86) | 1.9 (0.84)
  Q9, AUC At Day 29: number analyzed (Participants) | 95 | 92 | 91 | 91
  Q9, AUC At Day 29 | 2.7 (1.00) | 2.9 (0.84) | 2.7 (0.96) | 2.1 (0.93)
  Q10, AUC At Day 1: number analyzed (Participants) | 86 | 87 | 91 | 88
  Q10, AUC At Day 1 | 2.8 (0.82) | 2.7 (0.69) | 2.7 (0.85) | 2.2 (0.95)
  Q10, AUC At Day 29: number analyzed (Participants) | 84 | 84 | 88 | 86
  Q10, AUC At Day 29 | 2.9 (0.96) | 3.1 (0.77) | 2.9 (0.91) | 2.3 (0.93)
  Q11, AUC At Day 1: number analyzed (Participants) | 93 | 95 | 95 | 95
  Q11, AUC At Day 1 | 2.6 (0.89) | 2.6 (0.81) | 2.5 (0.89) | 2.0 (0.89)
  Q11, AUC At Day 29: number analyzed (Participants) | 94 | 92 | 91 | 91
  Q11, AUC At Day 29 | 2.8 (0.92) | 2.9 (0.85) | 2.8 (0.95) | 2.2 (0.92)
  Q12, AUC At Day 1: number analyzed (Participants) | 82 | 90 | 78 | 69
  Q12, AUC At Day 1 | 2.2 (0.96) | 2.3 (0.79) | 2.2 (0.87) | 1.8 (0.96)
  Q12, AUC At Day 29: number analyzed (Participants) | 81 | 85 | 84 | 78
  Q12, AUC At Day 29 | 2.4 (1.06) | 2.6 (0.90) | 2.4 (1.01) | 1.8 (0.86)

ADVERSE EVENTS:
Time Frame: Approximately 29 days
Arm/Group | OralBalance Moisturizing Gel | Oral Rinse | Moisturizing Mouth Spray | Water Only Use
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/98 | 0/98 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/101 | 1/98 | 2/98 | 0/99
Other Adverse Events (participants affected / at risk) | 17/101 | 21/98 | 12/98 | 20/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OralBalance Moisturizing Gel (N=101) | Oral Rinse (N=98) | Moisturizing Mouth Spray (N=98) | Water Only Use (N=99)
CARDIAC ARREST (Cardiac disorders) | 0 | 1 | 0 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 1 | 0
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OralBalance Moisturizing Gel (N=101) | Oral Rinse (N=98) | Moisturizing Mouth Spray (N=98) | Water Only Use (N=99)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 0
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Tongue Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
MOUTH INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
LIP INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OROPHARYNGAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
ORAL HERPES (Infections and infestations) | 2 | 1 | 0 | 3
BRONCHITIS (Infections and infestations) | 1 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 3 | 1 | 1
HORDEOLUM (Infections and infestations) | 0 | 1 | 0 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1
LARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 1
DEVICE EXPULSION (General disorders) | 1 | 0 | 0 | 0
APPLICATION SITE ANAESTHESIA (General disorders) | 0 | 1 | 0 | 0
PAIN (General disorders) | 0 | 0 | 1 | 0
PRODUCT TASTE ABNORMAL (General disorders) | 0 | 0 | 1 | 0
APPLICATION SITE PAIN (General disorders) | 0 | 0 | 1 | 0
DEVICE FAILURE (General disorders) | 0 | 0 | 0 | 2
PARAESTHESIA ORAL (Gastrointestinal disorders) | 1 | 0 | 0 | 0
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
LIP DRY (Gastrointestinal disorders) | 1 | 0 | 0 | 0
CHEILITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 1 | 0
LIP EXFOLIATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GINGIVAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 1 | 1 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GLOSSODYNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GINGIVAL INFLAMMATION (Gastrointestinal disorders) | 0 | 1 | 0 | 1
TONGUE COATED (Gastrointestinal disorders) | 1 | 3 | 2 | 1
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 0 | 1 | 0 | 0
TONGUE DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ORAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 0 | 0 | 1
LIP ULCERATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.